CLINICAL TRIAL: NCT07116317
Title: Determination of the Relationship Between Orthodontic Malocclusion Severity and Salivary Cortisol, Dehydroepiandrosterone and Chromogranin A Levels
Brief Title: Salivary Stress Markers Associated With Malocclusion Severity
Status: Not yet recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: ortho04/2025
Record Dates: First submitted 2025-08-01; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Malocclusion
Keywords: malocclusion; stress; cortisol; Dehydroepiandrosterone; Chromogranin A
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Saliva samples will be stored until the day they are to be biochemically analyzed to prevent deterioration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with normal or minor malocclusion: Patients with a Dental Aesthetic Index score of ≤25
- Patients with moderate malocclusion: Patients with a Dental Aesthetic Index score of 26-30
- Patients with severe malocclusion: Patients with a Dental Aesthetic Index score of 31-35
- Patients with obstructive malocclusion: Patients with a Dental Aesthetic Index score of ≥36

SUMMARY:
The aim of this observational study is to evaluate the relationship between the severity of orthodontic malocclusion and psychophysiological stress levels in individuals aged 12 to 18 years. The study will investigate the association between malocclusion severity and both stress-related salivary biomarkers and psychosocial factors.

The primary research question is as follows:

As the severity of orthodontic malocclusion increases, do levels of salivary stress biomarkers (cortisol, DHEA, and chromogranin A), self-esteem, and social appearance anxiety significantly change in adolescent individuals?

Method:

The study will include participants between the ages of 12 and 18. The severity of malocclusion will be assessed through clinical examination. Psychological assessments will be conducted using structured questionnaires to measure self-esteem and social appearance anxiety. In addition, saliva samples collected in the morning will be analyzed using the ELISA method to determine levels of cortisol, DHEA, and chromogranin A (CgA). The data will be statistically analyzed to identify the potential relationship between orthodontic malocclusion and biological and psychosocial indicators of stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12 and 18,
* Patients with all permanent teeth,
* Patients with the ability to read and understand,
* Patients with a cephalometric evaluation file and maxillary and mandibular impression dental models before diagnostic orthodontic treatment.

Exclusion Criteria:

* Presence of any congenital craniofacial deformity (cleft lip and palate or any other craniofacial syndrome or deformity),
* Patients who have previously initiated or completed orthodontic treatment,
* Patients with a history of psychiatric illness, the presence of caries, facial asymmetry, and any skin deformity affecting facial aesthetics.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients coming to Recep Tayyip Erdogan University Faculty of Dentistry Orthodontics Clinic for routine orthodontic treatment
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale Score | First day
  A four-point scale will be used to score responses to the 10 items. Positive questions are scored as 3: Strongly agree; 2: Agree; 1: Disagree; and 0: Strongly disagree, while negative questions are scored as 0: Strongly agree; 1: Agree; 2: Disagree; and 3: Strongly disagree. According to the final total score of the Rosenberg Self-Esteem Scale scores between 0-15, 15-25, and 25-30 indicate low, normal, and high self-esteem levels, respectively.
Social Appearance Anxiety Scale Score | First day
  Social Appearance Anxiety Scale 16-item scale concerns how patients feel about their appearance. A score of 1 to 5 is given for each item as follows: 1, completely disagree; 2, partially disagree; 3, unsure; 4, partially agree; 5, I completely agree. Scores range from 16 to 80, with higher scores representing greater social appearance anxiety.
Collection of Saliva Samples | Second day
  Prior to saliva collection, participants will be instructed to abstain from caffeine and/or nicotine for at least 4 hours and alcohol for at least 24 hours. Saliva will be collected between 9:00 AM and 11:00 AM to minimize circadian variations. Unstimulated saliva flow rate will be collected over 10 minutes using the spitting method and will be expressed in mL/min.

SECONDARY OUTCOMES:
Concentration of Cortisol, Dehydroepiandrosterone (DHEA) and Chromogranin A | approximately in the 4th month
  Salivary cortisol, DHEA and Chromogranin A will be obtained from unstimulated whole saliva samples. Saliva samples will be stored at -20°C until analyzed. Human salivary cortisol, DHEA, and Chromogranin A will be measured using radioenzyme immunoassay using a commercial enzyme-linked immunosorbent assay (ELISA) kit according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Oguz KOSE, Professor Dr., Study Director — Recep Tayyip Erdogan University Faculty of Dentistry
Locations (1):
- Department of Orthodontics of the Faculty of Dentistry of Recep Tayyip Erdogan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No